CLINICAL TRIAL: NCT05110768
Title: A Randomized, Placebo-controlled Study of the Treatment of Iron Deficiency Anemia (IDA) by Ferric Pyrophosphate Citrate (FPC) Delivered Via Infusion Pump in Patients Receiving Home Infusion Therapy
Brief Title: Treatment of (IDA) by (FPC) Delivered Via Infusion Pump in Patients Receiving Home Infusion Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-HI-01
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Iron Deficiency Anemia
Keywords: Ferric Pyrophosphate Citrate
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FPC 20 mg Fe IV by infusion over 12 hours every other day (Experimental): Patients in the FPC arm will receive FPC 20 mg Fe IV by infusion over 12 hours every other day (qOD), for a total duration of up to 12 weeks plus a one-week follow-up after the last study drug treatment.For patients whose duration of therapy is >10 hours, patients will receive a 12-hour infusion of FPC.
  Interventions: Drug: Triferic AVNU
- Placebo (Placebo Comparator): Patients in the placebo arms will receive IV placebo on the same schedule for 12 weeks. All patients are eligible to receive Rescue conventional IV iron if criteria are met and the patient's principal physician agrees.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Triferic AVNU — Triferic AVNU is an iron salt that is approved for the maintenance of Hgb in chronic kidney disease patients on hemodialysis. It is experimental in this study because it has not yet been approved for patients receiving home infusion therapy
  Other Names: Ferric Pyrophosphate Citrate (FPC)
  Arms: FPC 20 mg Fe IV by infusion over 12 hours every other day
Other: Placebo — normal TPN solution without FPC on alternate days with TPN supplemented with multivitamins.
  Arms: Placebo

SUMMARY:
The main purpose is to determine whether FPC, administered via infusion, is safe and effective for the treatment of iron deficiency anemia (IDA) in patients receiving Home Infusion therapies (HI).

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo-controlled, multi-center, clinical trial of the safety and efficacy of FPC infusion for patients diagnosed with IDA receiving therapy home infusion therapy. The study will be open label placebo-controlled using an objective endpoint (Hgb). A total of 75 home infusion patients will be enrolled.

Subjects will be randomized to receive FPC starting at Day 1; Patients in the FPC arm will receive FPC 20 mg Fe IV by infusion over 12 hours every other day (qOD), for a total duration of up to 12 weeks plus a one-week follow-up after the last study drug treatment. For patients whose duration of therapy is >10 hours, patients will receive a 12-hour infusion of FPC. Patients in the placebo arms will receive IV placebo on the same schedule for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Receiving a home infusion therapy requiring IV administration of fluid via an indwelling access device for up to 12 hours daily, 7 days a week, for >4 weeks
* Diagnosed with Iron deficiency anemia (Hgb <11.5 g/dL Female and <12 g/dL Male)
* CHr <29 pg./mL
* Serum Ferritin <100 ng/mL
* TSAT <20%
* Ability and willingness to adhere to the home infusion administration of FPC/Placebo.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

* Use of oral or intravenous iron within 4 weeks prior to randomization.
* Pregnancy or lactation
* Any febrile illness (oral temperature > 100.4°F, 38°C) during screening.
* Treatment with another investigational drug within 30 days of Randomization
* Current smoker or tobacco use within ≥3 months
* Known cause of anemia other than iron deficiency (e.g., sickle cell disease, thalassemia, pure red cell aplasia, hemolytic anemia, myelodysplastic syndrome, Vitamin B12 deficiency …etc.)
* Vitamin deficiency at Screening Visit
* Iron overload that contraindicates further iron supplementation as deemed by the PI.
* Prior documented hypersensitivity reaction (anaphylaxis) to IV iron administration
* History of drug or alcohol abuse within the last 6 months.
* Known active tuberculosis, fungal, viral, or parasitic infection requiring anti-microbial therapy or anticipated to require anti-microbial therapy during the patient's participation in this study.
* Known positive status for hepatitis B surface antigen (hepatitis B testing is not required as part of this protocol).
* Known human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this protocol).
* Cirrhosis of the liver based on histological criteria or clinical criteria (e.g., presence of ascites, esophageal varices, spider nevi, or history of hepatic encephalopathy).
* Hepatitis C infection if ALT and/or AST levels are consistently greater than twice the upper limit of normal at any time during the 2 months prior to randomization.
* Subjects who are anticipated to be unable to complete the entire study (e.g., due to a concurrent disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
The efficacy of FPC in treating Iron deficiency anemia (IDA) by FPC infusion in patients receiving Home Infusion therapies (HI). | Change from Baseline in serum iron at 17 weeks
  The efficacy will be done by assessing the change from baseline in serum iron to end of treatment (EoT). EoT is defined as the average of the last 2 bi-weekly Hgb values obtained at end of study or if the patient is prematurely terminated for any reason.

SECONDARY OUTCOMES:
The proportion of "patient responders," | Change from Baseline in HgB at 17 weeks.
  ≥ 1 g/dL increase from baseline in Hgb.
Iron delivery to the erythron. | Change from Baseline in CHr and sTfR levels at 17 weeks
  estimated by change in serum reticulocyte count, reticulocyte hemoglobin (CHr) and soluble transferrin receptor (sTfR) levels.
Need for rescue therapy | up to 17 weeks
  The number of patients requiring oral iron, intravenous iron and/or blood /packed RBC transfusions and the amount of intravenous iron and blood/packed cell transfusions.
Treatment (Patient) failure. | up to 17 weeks
  Incidence and time to development of iron deficiency defined as serum ferritin < 100 µg/L and TSAT< 20% confirmed by a consecutive repeat value (any time ≥ 1 day and ≤ 2 weeks after the first value).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical

IPD SHARING:
Plan to Share IPD: Yes